CLINICAL TRIAL: NCT00307580
Title: Cathflo Activase (Alteplase) Pediatric Study (CAPS)
Brief Title: Cathflo Activase Pediatric Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A2404g
Record Dates: First submitted 2006-03-25; First posted 2006-03-28 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Dysfunctional Central Venous Access Devices (CVADS)
Keywords: CVADS
MeSH Terms: interventions — Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Cathflo Activase (Alteplase)

SUMMARY:
This was a Phase IV, open-label, single-arm, multicenter trial that was to be conducted at ~60 sites in the United States. Approximately 300 pediatric subjects with dysfunctional CVADs (including catheters with valves, multiple lumens, umbilical catheters, and implanted ports) were to be treated with up to two serially instilled doses of Cathflo Activase.

ELIGIBILITY:
Inclusion Criteria:

Subjects had to meet the following inclusion criteria to be eligible for study entry:

* Less than 17 years of age
* Clinically stable
* Occlusion of CVAD (including catheters with valves, multiple lumens, umbilical catheters, and implanted ports)
* For subjects who weighed >= 10 kg, inability to withdraw 3 mL of blood from the CVAD
* For subjects who weighed < 10 kg, inability to withdraw 1 mL of blood from the CVAD
* Ability to infuse fluids at the volume necessary to instill Cathflo Activase into the CVAD
* Written informed consent and assent (if appropriate) provided by parent or legal guardian and compliance with study assessments for the full duration of the study

Exclusion Criteria:

* Ability to withdraw blood following subject repositioning
* CVAD insertion < 48 hours prior to enrollment
* Selected study catheter implanted specifically for hemodialysis
* Evidence of mechanical, non-thrombotic occlusion of the CVAD (e.g., kink in the CVAD or suture constricting the catheter)
* Previous enrollment in this study
* Use of fibrinolytic agent (e.g., alteplase, reteplase, tenecteplase, urokinase, streptokinase) within 24 hours of enrollment
* At high risk for bleeding events, embolic complications (i.e., recent pulmonary embolism, deep vein thrombosis, endarterectomy, clinically significant right-to-left shunt) in the opinion of the investigator, or with known condition for which bleeding constituted a significant hazard
* Known hypersensitivity to alteplase or any component of the formulation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300
Dates: Start 2002-04; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, as measured by the incidence of intracranial hemorrhage during the treatment with Cathflo Activase, in restoring function to dysfunctional CVADs in pediatric populations.

SECONDARY OUTCOMES:
To estimate the rate of restoration of function to dysfunctional CVADs following administration of up to two instillations of Cathflo Activase.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Blaney, PharmD, Study Director — Genentech, Inc.